CLINICAL TRIAL: NCT03232840
Title: Evaluation of an E-learning to Prevent Wrong Site Surgery in Anesthesia.
Brief Title: E-learning to Prevent Wrong Site Surgery in Anesthesia
Acronym: ELPSite
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0228
Record Dates: First submitted 2017-07-05; First posted 2017-07-28 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-10

CONDITIONS: Medical Errors : Wrong Site Surgery in Regional Anesthesia
Keywords: wrong site surgery in regional anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this observational study is to assess the efficiency of an e-learning in order to put into practice some preventive measures to avoid wrong site surgery during anesthesia.

DETAILED DESCRIPTION:
Before the study, the investigators selected 7 preventive measures to avoid wrong site surgery during regional anesthesia combined or not with general anesthesia . These measures were learned to the entire anesthesia team (nurse, resident and anesthesiologist) during conventional meetings. An initial evaluation of the application of these measures will be carried out before the introduction of e-learning. This assessment will be conducted by nurses without the knowledge of the anesthetic team evaluated. After this initial evaluation, e-learning will be broadcast on the hospital intranet. Then a second evaluation of the application of the preventive measures will be carried out 6 month and 1 year after the introduction of e-learning.

ELIGIBILITY:
Inclusion criteria:

* patient undergoing regional anesthesia with or without general anesthesia

Exclusion criteria:

* general anesthesia without regional anesthesia
* perimedullar anesthesia
* bilateral surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing anesthesia in Lapeyronie Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the application of each of the 7 preventive measures using a questionnaire filled by a nurse not involved in the regional anesthesia procedure | 1 day
  Evaluation of the application of each of the 7 preventive measures using a questionnaire filled by a nurse not involved in the regional anesthesia procedure. This questionnaire simply indicates whether a measure has been applied or not

OTHER OUTCOMES:
Assessment of the application of each of the 7 preventive measures according to various clinical parameters | 1 day
  Evaluation of the application of each of the 7 preventive measures according to the clinical parameters of the patients followed (age of the patient, ASA physical status, type of surgery, type of anesthesia, period of the day or week, Emergency or elective).
Evaluation of the application of the preventive measures following the introduction of the e-learning in the anesthesia team. | 6 month and 1 year
  Evaluation of the application of the preventive measures following the introduction of the e-learning in the anesthesia team.

CONTACTS AND LOCATIONS:
Overall Officials: BIBOULET Philippe, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC